CLINICAL TRIAL: NCT04319302
Title: Isolated Vascularized Gastric Tube Biliary Enteric Drainage: A Paediatric Case Series Experience.
Status: Completed | Type: Observational
Sponsor: University of KwaZulu (Other)
Responsible Party: Principal Investigator, Hansraj Mangray, Head of Paediatric Surgery, Greys Hospital, University of KwaZulu
Other Study IDs: C3619112712050
Record Dates: First submitted 2020-03-19; First posted 2020-03-24 (Actual); Last update posted 2020-03-30 (Actual); Status verified 2020-03

CONDITIONS: Biliary Obstruction; Choledochal Cyst
Keywords: Choledochal cyst; Paediatric; Roux-en-Y; Bile drainage; Gastric conduit
MeSH Terms: conditions — Choledochal Cyst | interventions — Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Paediatric biliary obstruction: This was a retrospective review of all paediatric patients who had undergone an IVGT graft procedure for biliary tract anatomical obstruction in the past five years. We looked at the indications for surgery, the demographic profile of the patients, outcomes following surgery and outlined the surgical technique used.
  Interventions: Procedure: Isolated Vascularized Gastric Tube (IVGT) graft

INTERVENTIONS:
Procedure: Isolated Vascularized Gastric Tube (IVGT) graft — A conduit was created by tubularising a vascularized segment of the greater curve of the antrum of the stomach and this was used between the remaining common hepatic duct and the duodenum.

SUMMARY:
This was a retrospective case series experience of paediatric patients who had an Isolated vascularized gastric tube biliary enteric drainage procedure for biliary obstruction over the past five years. We reviewed our experience and outcomes.

DETAILED DESCRIPTION:
Background

Despite the enormous surgical advancements in the last century, access to the biliary system is lost when a Roux-en-Y (RY) biliary drainage procedure is performed. Attempts have been made to overcome this inconvenient sequel of RY biliary drainage by the use of variations in the RY anastomosis, small bowel grafts and vascular grafts. These have been predominantly unsuccessful. The use of an Isolated Vascularized Gastric Tube (IVGT) graft has been reported in the literature, and this was successfully used for adult patients with common bile duct injuries. The investigators have adopted the technique of using an IVGT graft for bile duct reconstruction in the paediatric patients at their institution.

Method

The investigators reviewed theirr experience at Greys Hospital, Pietermaritzburg. This was a retrospective review of all paediatric patients who had undergone an IVGT graft procedure for biliary tract anatomical obstruction in the past five years. The investgators looked at the indications for surgery, the demographic profile of the patients, outcomes following surgery and outlined the surgical technique used.

ELIGIBILITY:
Inclusion Criteria:

* All patients from birth to 12 years with biliary tract obstruction requiring surgery.

Exclusion Criteria:

* biliary atresia

Max Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: This was a retrospective review of all paediatric patients at Greys Hospital who had undergone an IVGT graft procedure for biliary tract anatomical obstruction in the past five years
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2005-01 (Actual); Primary Completion 2020-01 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
Bile drainage | 30 days
  Effectiveness of procedure to allow drainage of bile into the bowel.

SECONDARY OUTCOMES:
Complications of procedure | 30 days
  What complications were encountered following the procedure

OTHER OUTCOMES:
Complications | 1 year
  What were the long term complications

CONTACTS AND LOCATIONS:
Locations (1):
- Greys Hospital, Pietermaritzburg, KwaZulu-Natal, South Africa

IPD SHARING:
Plan to Share IPD: No
Data will be retained by researchers and ade available on request.